CLINICAL TRIAL: NCT00550836
Title: Randomized Phase II Trial of Panitumumab, Erlotinib and Gemcitabine vs. Erlotinib and Gemcitabine in Patients With Untreated, Metastatic Pancreatic Adenocarcinoma
Brief Title: Erlotinib and Gemcitabine With or Without Panitumumab in Treating Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N064B; NCI-2009-01089 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000571863 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-10-26; First posted 2007-10-30 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-02

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; duct cell adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Panitumumab; Erlotinib Hydrochloride; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: GE (Active Comparator): Patients receive 1000 mg/m^2 gemcitabine hydrochloride IV on days 1, 8, and 15; and 100 mg oral erlotinib hydrochloride on days 1-28. Treatment repeats every 28 days for 2 courses. Patients achieving a complete response (CR) after 2 courses receive 2 additional courses of treatment; patients achieving a partial response (PR) receive retreatment as above. Patients achieving a CR after 4 courses of treatment receive erlotinib hydrochloride until the first disease progression. After the first progression, patients are retreated with gemcitabine hydrochloride and erlotinib hydrochloride until second progression.
  Interventions: Drug: erlotinib hydrochloride; Drug: gemcitabine hydrochloride
- Arm B: PGE (Experimental): Patients receive 1000 mg/m^2 gemcitabine hydrochloride IV on days 1, 8, and 15; 100 mg oral erlotinib hydrochloride on days 1 - 28; and 4.0 mg/kg panitumumab IV on days 1 and 15. Treatment repeats every 28 days for 2 courses. Patients achieving a CR after 2 courses receive 2 additional courses of treatment; patients achieving a PR receive retreatment as above. Patients achieving a CR after 4 courses of treatment receive erlotinib hydrochloride and panitumumab until the first disease progression. After the first progression, patients are retreated with gemcitabine hydrochloride, erlotinib hydrochloride, and panitumumab until second progression.
  Interventions: Biological: panitumumab; Drug: erlotinib hydrochloride; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Biological: panitumumab — Given IV
  Arms: Arm B: PGE
Drug: erlotinib hydrochloride — Given orally
Drug: gemcitabine hydrochloride — Given IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as panitumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Panitumumab may also stop the growth of pancreatic cancer by blocking blood flow to the tumor.

PURPOSE: This randomized phase II trial is studying how well giving panitumumab together with gemcitabine and erlotinib works compared to giving gemcitabine and erlotinib alone in treating patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess whether the addition of panitumumab (a dual-epidermal growth factor receptor inhibitor) to standard chemotherapy comprising gemcitabine hydrochloride and erlotinib hydrochloride results in an improvement in overall survival of patients with previously untreated, metastatic adenocarcinoma of the pancreas.

Secondary

* To compare objective response rates, progression-free survival, time to treatment failure, quality of life, and adverse event rates in patients treated with these regimens.
* To evaluate the downstream marker, KRAS, in stool specimens.

OUTLINE: This is a multicenter study. Patients are stratified according to ECOG performance status (0 vs 1) and prior adjuvant chemotherapy (yes vs no). The first 6 patients are assigned to arm II. Subsequent patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15 and oral erlotinib hydrochloride once daily on days 1-28. Treatment repeats every 28 days for 2 courses. Patients achieving a complete response (CR) after 2 courses receive 2 additional courses of treatment; patients achieving a partial response (PR) receive retreatment as above in the absence of disease progression or unacceptable toxicity. Patients achieving a CR after 4 courses of treatment receive maintenance therapy comprising erlotinib hydrochloride daily until the first disease progression. After the first progression, patients are retreated with gemcitabine hydrochloride and erlotinib hydrochloride until second progression (using the first progression tumor measurements as the new baseline reference).
* Arm II: Patients receive gemcitabine hydrochloride and erlotinib hydrochloride as in arm I and panitumumab IV over 1 hour on days 1 and 15. Treatment repeats every 28 days for 2 courses. Patients achieving a CR after 2 courses receive 2 additional courses of treatment; patients achieving a PR receive retreatment as above in the absence of disease progression or unacceptable toxicity. Patients achieving a CR after 4 courses of treatment receive maintenance therapy comprising erlotinib hydrochloride daily and panitumumab every 2 weeks until the first disease progression. After the first progression, patients are retreated with gemcitabine hydrochloride, erlotinib hydrochloride, and panitumumab until second progression (using the first progression tumor measurements as the new baseline reference).

Stool samples are collected at baseline and analyzed for KRAS mutations via protein analyses.

Quality of life will be assessed at baseline, every 2 courses during treatment, and at the end of treatment.

After the second progression, patients are followed every 3-6 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas (ductal or undifferentiated)

  * Metastatic disease
* No islet cell, acinar cell, or cystadenocarcinomas
* No locally advanced disease
* No history or known presence of CNS metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 3 months
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Total bilirubin ≤ 2 times upper limit of normal (ULN) (patients may be stented)
* AST ≤ 2.5 times ULN
* Creatinine ≤ 2.0 times ULN
* Magnesium ≥ lower limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Willing to provide a stool specimen
* No malignancy diagnosed within the past 3 years except basal cell or squamous cell skin cancer, prostate cancer (Gleason < 7), or carcinoma in situ of the cervix
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements
* No clinically significant cardiovascular disease (i.e., myocardial infarction, unstable angina, symptomatic congestive heart failure, or serious uncontrolled cardiac arrhythmia) within the past year
* No known positive test(s) for HIV infection, hepatitis C virus, or acute or chronic active hepatitis B infection
* No liver dysfunction from cirrhosis or viral hepatitis
* No enteral hyperalimentation
* No grapefruit or grapefruit juice during the study

PRIOR CONCURRENT THERAPY:

* Recovered from prior therapy
* More than 4 months since prior radiotherapy, immunotherapy, or biologic therapy
* More than 4 weeks since prior and no elective or planned major surgery
* More than 2 weeks since prior minor and no elective or planned surgery
* No prior cytotoxic chemotherapy for metastatic disease

  * Adjuvant chemotherapy for completely resected disease or chemoradiotherapy for locally advanced disease is allowed, provided it was administered > 6 months prior to study entry

    * Adjuvant chemotherapy must not have contained an EGFR inhibitor
  * Gemcitabine hydrochloride used as either a radiosensitizer or as maintenance therapy is allowed, provided more than 6 months have elapsed since the last day of treatment
* No prior anti-EGFR antibody therapy (e.g., cetuximab) or treatment with small molecule EGFR inhibitors (e.g., gefitinib hydrochloride, erlotinib hydrochloride, or lapatinib)
* No concurrent immunotherapy or radiotherapy
* No other concurrent chemotherapy
* No concurrent colony-stimulating factors during the first course of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-03; Primary Completion 2010-11 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George P. Kim, MD, Study Chair — Mayo Clinic
Locations (262):
- United States (262):
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Pacific Cancer Institute - Maui, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Ochsner Health Center - Bluebonnet, Baton Rouge, Louisiana
  - Ochsner Health Center - Covington, Covington, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria, Minnesota
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls Medical Group, PA, Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Luther Midlelfort Hospital, Eau Claire, Wisconsin
  - Midelfort Clinic - Luther, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Derived] Halfdanarson TR, Foster NR, Kim GP, Meyers JP, Smyrk TC, McCullough AE, Ames MM, Jaffe JP, Alberts SR. A Phase II Randomized Trial of Panitumumab, Erlotinib, and Gemcitabine Versus Erlotinib and Gemcitabine in Patients with Untreated, Metastatic Pancreatic Adenocarcinoma: North Central Cancer Treatment Group Trial N064B (Alliance). Oncologist. 2019 May;24(5):589-e160. doi: 10.1634/theoncologist.2018-0878. Epub 2019 Jan 24. PMID 30679315

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: GE | Arm B: PGE
Started | 49 | 55
Completed | 46 | 46
Not Completed | 3 | 9
Not completed — Withdrawal by Subject | 3 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: GE | Arm B: PGE | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Continuous [Median (Full Range); unit: years] | 60.5 [37 to 81] | 62 [37 to 79] | 61.5 [37 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 29 | 31 | 60
Region of Enrollment [Number; unit: participants]
  United States | 46 | 46 | 92

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall Survival is defined as the time from registration to death due to any cause. The estimate will be done using the Kaplan-Meier method. The primary goal of this trial is to compare the experimental arm (Arm B) to the standard arm (Arm A). The primary analysis will be a comparison of Arm A to Arm B using a one-sided log-rank test between the 2 Kaplan-Meier curves.
Time Frame: Up to 2 years
Population: All treated patients that were eligible were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: GE | Arm B: PGE
Number analyzed (Participants) | 46 | 46
months | 4.2 [3.5 to 7.8] | 8.3 [4.5 to 10]
Statistical Analysis 1: Comparison: Arm A: GE vs Arm B: PGE; It was calculated that 39 participants randomized in a 1:1 fashion between the 2 arms would have 80% to detect a difference in median survival of 6 vs. 9.7 months for GE vs. PGE respectively with a minimum follow up of 6 months. Sample size was determined using a 1-sided log-rank test at alpha=0.20; Test type: Superiority; p = 0.36, Log Rank

2. Secondary Outcome: Confirmed Response Rate
Description: Evaluated using RECIST version 1.0. Confirmed tumor response rate was defined as achieving partial response (PR) or complete response (CR) in two consecutive assessments at least 6 weeks apart. CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. The confirmed response rate is reported as the number of participants with confirmed responses divided by the number of evaluated participants.
Time Frame: Up to 2 years
Population: All patients that started protocol treatment and were evaluated were included in this analysis.
Measure: Number (95% Confidence Interval); unit: rate of confirmed response
Arm/Group | Arm A: GE | Arm B: PGE
Number analyzed (Participants) | 46 | 46
rate of confirmed response | 0.087 [0.024 to 0.208] | 0.065 [0.014 to 0.179]
Statistical Analysis 1: Comparison: Arm A: GE vs Arm B: PGE; Test type: Other; p = 1.0, Fisher Exact

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the time from randomization to documentation of disease progression or death, whichever comes first. Progression is defined as at least a 20% increase in the sum of longest dimension (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. The distribution of progression-free survival will be estimated using the method of Kaplan-Meier. The progression-free survival curves will be compared between the 2 arms using a log-rank test.
Time Frame: Up to 2 years
Population: All treated patients were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: GE | Arm B: PGE
Number analyzed (Participants) | 46 | 46
months | 2.0 [1.8 to 3.3] | 3.6 [2.3 to 4.5]
Statistical Analysis 1: Comparison: Arm A: GE vs Arm B: PGE; Test type: Superiority; p = 0.419, Log Rank

4. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined to be the time from the date of randomization to the date at which the patient is removed from treatment due to progression, adverse events, or refusal. If the patient is considered to be a major treatment violation or is taken off study as a nonprotocol failure, the patient will be censored on the date they are removed from treatment. The time to treatment failure will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 2 years
Population: All eligible treated patients were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: GE | Arm B: PGE
Number analyzed (Participants) | 46 | 46
months | 2.0 [1.8 to 2.5] | 3.8 [2.0 to 4.2]
Statistical Analysis 1: Comparison: Arm A: GE vs Arm B: PGE; Test type: Other; p = 0.36, Log Rank

5. Secondary Outcome: Frequency and Severity of Observed Adverse Effects
Description: Patients are assessed for Adverse events each cycle using the Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0). The maximum grade for each type of adverse event will be recorded for each patient, and tables will be reviewed to determine adverse event patterns. The number of patients in each arm that reported a grade 3 or higher adverse event and a grade 4 or higher adverse event are reported.
  A complete listing of all adverse events is reported in the Adverse Events section.
Time Frame: Up to 2 years
Population: All evaluable patients were included in this analysis.
Measure: Number; unit: participants
Arm/Group | Arm A: GE | Arm B: PGE
Number analyzed (Participants) | 46 | 46
participants
  Grade 3+ Adverse Event | 41 | 41
  Grade 4+ Adverse Event | 15 | 14

ADVERSE EVENTS:
Arm/Group | Arm A: GE | Arm B: PGE
Serious Adverse Events (participants affected / at risk) | 30/46 | 27/46
Other Adverse Events (participants affected / at risk) | 45/46 | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: GE (N=46) | Arm B: PGE (N=46)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 6 (6) | 6 (6)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 2 (2)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 2 (2)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Jejunal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (10) | 3 (4)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 9 (9) | 4 (4)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2)
Disease progression (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 5 (5) | 4 (4)
Fever (General disorders) | 2 (2) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Gallbladder infection (Infections and infestations) | 1 (1) | 0 (0)
Infectious colitis (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 3 (4) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Bilirubin increased (Investigations) | 4 (4) | 3 (3)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 3 (3) | 2 (2)
Weight loss (Investigations) | 2 (2) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (4) | 2 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 9 (9) | 6 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: GE (N=46) | Arm B: PGE (N=46)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 8 (11) | 10 (21)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (8) | 5 (6)
Ascites (Gastrointestinal disorders) | 1 (1) | 4 (4)
Constipation (Gastrointestinal disorders) | 5 (13) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 25 (47) | 24 (60)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 30 (64) | 35 (79)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 13 (21) | 22 (32)
Chest pain (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 4 (7)
Fatigue (General disorders) | 15 (25) | 19 (44)
Fever (General disorders) | 1 (1) | 3 (3)
Pain (General disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Gingival infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (3)
Nail infection (Infections and infestations) | 0 (0) | 1 (2)
Paranasal sinus infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 4 (4)
Vaginal infection (Infections and infestations) | 1 (2) | 0 (0)
Venous injury - Extremity-upper (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 10 (12) | 7 (13)
Alkaline phosphatase increased (Investigations) | 11 (15) | 10 (12)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 10 (10)
Bilirubin increased (Investigations) | 3 (3) | 5 (6)
Cardiac troponin T increased (Investigations) | 0 (0) | 1 (1)
Coagulopathy (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 1 (2)
Laboratory test abnormal (Investigations) | 0 (0) | 2 (2)
Leukocyte count decreased (Investigations) | 7 (13) | 5 (7)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (5) | 2 (9)
Neutrophil count decreased (Investigations) | 25 (69) | 21 (45)
Platelet count decreased (Investigations) | 32 (95) | 29 (73)
Weight loss (Investigations) | 4 (7) | 5 (12)
Anorexia (Metabolism and nutrition disorders) | 12 (16) | 17 (30)
Blood glucose increased (Metabolism and nutrition disorders) | 3 (3) | 7 (9)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2) | 10 (17)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1) | 7 (13)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 5 (8) | 31 (102)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Serum sodium decreased (Metabolism and nutrition disorders) | 4 (7) | 3 (4)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mini mental status examination abnormal (Nervous system disorders) | 0 (0) | 1 (1)
Taste alteration (Nervous system disorders) | 3 (3) | 3 (5)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (22) | 12 (15)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (19) | 14 (25)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (11)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (7)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 5 (10) | 6 (20)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (22) | 31 (78)
Rash desquamating (Skin and subcutaneous tissue disorders) | 32 (90) | 43 (183)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Phlebitis (Vascular disorders) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 3 (3) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less